CLINICAL TRIAL: NCT02019966
Title: A Korean Cohort Study of TDF Rescue Therapy for Difficult-to-treat CHB Patients: a Comparison Between TDF Monotherapy and TDF-based Combination Therapy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0704
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: The Difficult-to-treat Chronic Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TDF monotherapy: TDF monotherapy - treated by tenofovir alone
  patients with CHB receiving rescue TDF (300mg once daily) monotherapy
- TDF-based combination therapy: TDF-based combination therapy - treated by tenofovir based combination therapy.
  patients with CHB receiving rescue TDF-based combination therapy (TDF 300mg once daily with any other nucleoside analogue such as lamivudine 100mg, telbivudine 600mg, or entecavir 1.0 mg once daily).

SUMMARY:
Antiviral resistance remains an important issue for long-term NA therapy. For lamivudine (LAM), the rtM204V/I and rtL180M mutations occur in more than 70% after 5 years of therapy. In Korea, primarily owing to limited subsidization policy in the health insurance system, many patients with LMV-resistance had been treated with either rescue ADV or ETV 1.0 mg monotherapy, ultimately leading to the higher prevalence of MDR strain. For those patients, rescue therapies of combining ADV with either ETV or LAM had been tried, but frequently with suboptimal responses. Rescue TDF monotherapy or TDF-based combination therapy are available in Korea for patients who had "difficult-to-treat" antiviral resistance owing to prior treatment failures. However, which is the better has not been evaluated yet. A long-term efficacy and safety of TDF-based rescue therapies in real practice for those patients should be necessary to revise the Korean guideline for the treatment of chronic hepatitis B in near future.

ELIGIBILITY:
Inclusion Criteria:

* more than 20 years old adults
* chronic hepatitis B
* the patients treated by tenofovir alone or tenofovir based combination therapy because of the previous treatment failure
* the patients who agree and singed on the consent form

Exclusion Criteria:

* co-infected patients with HCV, HDV or HIV
* pregnancy or breast feeding woman or female patients who are planning to be pregnant
* past history with hepatocellular carcinoma
* combined with other liver disease including wilson, alcoholic, NASH, alpha-1 antitrypsin deficiency liver disease.
* patients with hypersensitivity for drugs
* patients who were enrolled in other clinical study within 60 days
* patients who were eligible for the clinical study according to the investor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who had "difficult-to-treat" antiviral resistance owing to prior treatment failures
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who achieve a sustained HBV DNA < 60 IU/mL (Undetectable serum HBV DNA by PCR method) at each year during the on treatment follow-up period. | 1, 2, and 3 years after the treatment initiation.
  The viral response which is defined as serum HBV DNA < 60 IU/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Lim YS, Lee TH, Heo NY, Shim JH, Lee HC, Suh DJ. Entecavir plus adefovir combination treatment for chronic hepatitis B patients after failure of nucleoside/nucleotide analogues. Antivir Ther. 2012;17(1):53-60. doi: 10.3851/IMP1914. PMID 22267469
- [Background] van Bommel F, de Man RA, Wedemeyer H, Deterding K, Petersen J, Buggisch P, Erhardt A, Huppe D, Stein K, Trojan J, Sarrazin C, Bocher WO, Spengler U, Wasmuth HE, Reinders JG, Moller B, Rhode P, Feucht HH, Wiedenmann B, Berg T. Long-term efficacy of tenofovir monotherapy for hepatitis B virus-monoinfected patients after failure of nucleoside/nucleotide analogues. Hepatology. 2010 Jan;51(1):73-80. doi: 10.1002/hep.23246. PMID 19998272
- [Background] Tan J, Degertekin B, Wong SN, Husain M, Oberhelman K, Lok AS. Tenofovir monotherapy is effective in hepatitis B patients with antiviral treatment failure to adefovir in the absence of adefovir-resistant mutations. J Hepatol. 2008 Mar;48(3):391-8. doi: 10.1016/j.jhep.2007.09.020. Epub 2008 Jan 3. PMID 18199519
- [Background] Berg T, Marcellin P, Zoulim F, Moller B, Trinh H, Chan S, Suarez E, Lavocat F, Snow-Lampart A, Frederick D, Sorbel J, Borroto-Esoda K, Oldach D, Rousseau F. Tenofovir is effective alone or with emtricitabine in adefovir-treated patients with chronic-hepatitis B virus infection. Gastroenterology. 2010 Oct;139(4):1207-17. doi: 10.1053/j.gastro.2010.06.053. Epub 2010 Jun 20. PMID 20600025